CLINICAL TRIAL: NCT06488729
Title: Effectiveness of Foot Massage Applied Before a Bronchoscopy Procedure on Physiological Parameters and Anxiety: A Randomized Controlled Study
Brief Title: Foot Massage Applied Before a Bronchoscopy Procedure on Physiological Parameters and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Semra Aciksoz
Record Dates: First submitted 2024-05-31; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-04

CONDITIONS: Physiological Parameters; Anxiety; Bronchoscopy
Keywords: foot massage; anxiety; physiological parameters; bronchoscopy; randomized controlled trial
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The patients were separated into two groups with the randomisation method. These groups were named the foot massage group and the control group
Who Masked: Participant, Outcomes Assessor
Masking Description: To prevent interaction between groups, the data collection process of the control group was completed first.
  The researchers were not blinded to the groups, but the statistician was.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foot massage (Experimental): Foot massage was applied to the patients in the foot massage group.
  Interventions: Other: Foot massage
- Control (No Intervention): No procedures were applied to the control group other than clinical standard protocols.

INTERVENTIONS:
Other: Foot massage — Foot massage
  Arms: Foot massage

SUMMARY:
The goal of this randomized controlled trial is to assess the effectiveness of foot massage on physiological parameters and anxiety in patients undergoing bronchoscopy. The main questions it aims to answer are:

* Does foot massage applied before bronchoscopy affect physiological parameters?
* Does foot massage before bronchoscopy affect anxiety? Patients in the intervention group received foot massage once before bronchoscopy. Patients in the control group did not receive any treatment other than routine care.

DETAILED DESCRIPTION:
After the ethics committee and institutional permissions were obtained, patients scheduled for bronchoscopy were evaluated by the researcher for eligibility. First of all, they were informed about the study. Those who agreed to participate and delivered written consent were included in the sample. Individuals were assigned to the intervention and control groups by using block randomization. To prevent interaction between groups, the data collection process of the control group was completed first.A Personal Information Form, the State-Trait Anxiety Inventory, and a Vital Signs Monitoring Form were used to collect study data. In the control group, data were collected during the first arrival of the individuals (T1), 40 minutes after T1 (T2), and following bronchoscopy (T3). No procedures were applied to the control group other than clinical protocols. After the data collection process of the study was completed, the questions of the patients in the control group were answered.

The data of the intervention group were collected during the first arrival of the individuals (before the massage) (T1), 40 minutes after T1 (after the massage) (T2), and following bronchoscopy (T3).

Massage sessions lasted approximately 40 minutes, including 20 minutes for each foot.

ELIGIBILITY:
Inclusion Criteria:

aged ≥18 years communicate verbally be conscious no lesions on the feet or any problems that may affect the feet (diabetes, neurological disorder, etc.), no previous history of bronchoscopy no history of problems or anxiety no history of any disorder no acute pain no use of opioids or strong sedatives in the last week before recruitment to the study

Exclusion Criteria:

patients who underwent emergency bronchoscopy patients who do not want to participate in the research voluntarily

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2023-02-04 (Actual)

PRIMARY OUTCOMES:
physiological parameters | The data of the groups were collected during the first arrival of the individuals (before the massage), 40 minutes after the first measurement (after the massage), and following bronchoscopy.
  systolic blood pressure (mmHg)
physiological parameters | The data of the groups were collected during the first arrival of the individuals (before the massage), 40 minutes after the first measurement (after the massage), and following bronchoscopy.
  diastolic blood pressure (mmHg)
physiological parameters | The data of the groups were collected during the first arrival of the individuals (before the massage), 40 minutes after the first measurement (after the massage), and following bronchoscopy.
  heart rate (beats per minute (min-1 or bpm)
physiological parameters | The data of the groups were collected during the first arrival of the individuals (before the massage), 40 minutes after the first measurement (after the massage), and following bronchoscopy.
  respiratory rate (per minute)
physiological parameters | The data of the groups were collected during the first arrival of the individuals (before the massage), 40 minutes after the first measurement (after the massage), and following bronchoscopy.
  oxygen saturation (percent (%))
anxiety | The data of the groups were collected during the first arrival of the individuals (before the massage), 40 minutes after the first measurement (after the massage), and following bronchoscopy.
  The State Anxiety Inventory

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Turkey, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All information about the research can be shared
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2024-....